CLINICAL TRIAL: NCT06741826
Title: The Diagnostic Performance and Safety of Confocal Laser Endomicroscopy Guided Transbronchial Lung Cryobiopsy in the Diagnosis of Interstitial Lung Disease: a Randomised Controlled Trial
Brief Title: Confocal Laser Endomicroscopy Guided Cryobiopsy in the Diagnosis of Interstitial Lung Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Chief physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022YFC2404404-1
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group nCLE-NB-rEBUS (Experimental): According to the preoperative planning, the bronchoscope was placed at the bronchial opening of the target lobe segment, and the catheter was operated to reach the target lesion under the guidance of virtual navigation and after reaching the target lesion, the ultrasonic probe was opened to observe whether the ultrasonic image of the target lesion could be detected, and the image recording was collected to confirm that the virtual navigation catheter had accurately reached the target lesion. The ultrasound probe was removed, the TX ™ disposable transbronchoscopic dilator catheter was inserted to establish a working channel, and the nCLE was inserted to probe the benign and malignant status of the pleural lesion to determine the biopsy location and image recording was taken. Then the biopsy equipment was inserted and delivered to the target lesion for biopsy, and 5 pieces of biopsy tissue were collected.
  Interventions: Procedure: Navigation bronchoscopy combined with radial endobronchial ultrasound guided pulmonary nodule biopsy under needle-based confocal laser endomicroscopy.
- Group NB-rEBUS (Experimental): After anesthesia, electronic bronchoscope was inserted through laryngeal mask/tracheal intubation for routine bronchoscopy. According to the preoperative planning, the bronchoscope was placed at the bronchial opening of the target lobe segment, and the catheter was operated to reach the target lesion under the guidance of virtual navigation, and was placed about 1 cm away from the target. The radial ultrasonic probe was implanted, and after reaching the target lesion, the ultrasonic probe was opened to observe whether the ultrasonic image of the target lesion could be detected, and the image recording was collected to confirm that the virtual navigation catheter had accurately reached the target lesion. Take out the ultrasonic probe, insert it into the biopsy equipment, deliver it to the target lesion for biopsy, and collect 5 pieces of biopsy tissue.
  Interventions: Procedure: Navigation bronchoscopy combined with radial endobronchial ultrasound guided pulmonary nodule biopsy under needle-based confocal laser endomicroscopy.

INTERVENTIONS:
Procedure: Navigation bronchoscopy combined with radial endobronchial ultrasound guided pulmonary nodule biopsy under needle-based confocal laser endomicroscopy. — Navigation bronchoscopy combined with radial endobronchial ultrasound guided pulmonary nodule biopsy under needle-based confocal laser endomicroscopy.
  Other Names: Navigation bronchoscopy combined with radial endobronchial ultrasound guided pulmonary nodule biopsy.

SUMMARY:
A prospective multicenter randomized controlled trial was conducted to evaluate the diagnostic efficacy and safety of NCLE-NB-Rebus-guided peripheral pulmonary nodule biopsy, and to compare the diagnostic efficacy and safety of biopsy forceps biopsy and needle aspiration biopsy in peripheral pulmonary nodule biopsy guided by nCLE-NB-rEBUS.

DETAILED DESCRIPTION:
A prospective, multicenter, randomized controlled trial was conducted to evaluate the diagnostic efficacy and safety of nCLE-NB-rEBUS guided peripheral pulmonary nodule biopsy. Patients with peripheral pulmonary nodules suspected of lung cancer and pulmonary tuberculosis were enrolled to sign informed consent. Subjects were randomized to the nCLE-NB-rEBUS Group (Group A) or the NB-rEBUS Group (Group B) subgroup (1:1 ratio) according to the random number table, and subjects randomly assigned to Group A or Group B were again randomized to the biopsy forceps subgroup or biopsy needle subgroup by the random number table. The diagnostic efficacy and safety of the NCLE-NB-REbus group and the NB-rEBUS group were compared to evaluate whether nCLE could improve the diagnostic rate of NB-REbus-guided peripheral pulmonary nodule biopsy. The diagnostic efficacy and safety of using biopsy forceps and biopsy needle in peripheral pulmonary nodule biopsy guided by nCLE-NB-rEBUS were compared to determine the reasonable biopsy method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral pulmonary nodules suspected of lung cancer by CT examination
* Patients who intend to undergo a bronchoscopic lung biopsy to determine benign or malignant pulmonary nodules;
* Age ≥18 years
* Sign informed consent.

Exclusion Criteria:

* There is an uncorrectable coagulation disorder or anticoagulation therapy that cannot be stopped before surgery;
* Tumors can be seen in the bronchus
* Hemodynamic instability;
* Refractory hypoxemia;
* Patients with pregnant and lactating patients
* Any illness or condition that interferes with the completion of the initial or subsequent assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate of biopsy to obtain pathological diagnosis. | 6 months
  The biopsies obtained from the two groups were fixed in 10% formaldehyde and sent for pathological examination. The pathological diagnosis results were identified by two pathologists back to back, and the results were consistent, that is, confirmed. If the results are inconsistent, they will be identified by a third pathologist and finally determined by the three experts after discussion.

SECONDARY OUTCOMES:
Occurrence of operation-related complications | 6 months
  7 days of follow-up data (including bleeding, infection, pain, fever, etc.). Patients who did not obtain a confirmed diagnosis were followed up to 6 months after surgery to evaluate their diagnosis.

IPD SHARING:
Plan to Share IPD: No